CLINICAL TRIAL: NCT06051903
Title: Effect of Talar Mobilization With Movement Versus Acupuncture on Knee Pain and Function in the Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Kerolous Ishak Shehata, principle investigator, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: p.t.REC\012\004591
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Talar Mobilization Acupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Talar mobilization with movement (Experimental): (group A) postmenopausal women who receive the talar mobilization with movement technique for knee joint , their age raged from 50-60 years (n= 20)
  Interventions: Other: Mobilization wih movement
- Acupuncture for knee joint (Experimental): (group B) postmenopausal women who receive acupuncture for knee joint (n= 20), their age ranged from 50-60 years
  Interventions: Other: Mobilization wih movement

INTERVENTIONS:
Other: Mobilization wih movement — The purpose of this study is to determine the effect of talar mobilization with movement versus acupuncture on knee pain and function in the postmenopausal women

SUMMARY:
The purpose of this study is to determine the effect of talar mobilization with movement versus acupuncture on knee pain and function in the postmenopausal women

DETAILED DESCRIPTION:
A sample of forty postmenopausal women were selected from Department of Gynecology and Obstetrics, Participants were assigned into two groups (group A) postmenopausal women who receive the talar mobilization with movement technique for knee joint , their age raged from 50-60 years (n= 20) and (group B) postmenopausal women who receive acupuncture for knee joint (n= 20), their age ranged from 50-60 years and body mass index (BMI) for both groups were less than 30 kg/m2. All participants were evaluated through measuring knee range of motion by using goniometer and the degree of knee pain by using numeric rating scale and pressure algometer

ELIGIBILITY:
Inclusion Criteria:

* ) Females patients refered from orthopedic surgeon diagnosed with knee OA (2) Their age ranged from 50 _60 years old 3) Their BMI less than 30 kg/m2. 5) knee pain in the previous week with an intensity of at least 3 points on a numeric pain rating scale (NPRS ) (5) Patients limited ankle dorsiflexion ROM 6) All Patients had 3 points on NPS (7) Presence of knee pain for at least 3 moonths 8) All patients were given the arabic version of KOOS questionnaire

Exclusion Criteria:

* 1) Patients with Rheumatoid arthritis 2) Their BMI more than 30 kg/m2. 3) Unrelated to any traumatic knee event 4) Patients with Previous tibial fracture 5) Patients with Ankle instability 6) Patients with previous meniscal degeneration 7) Patients with hyper laxity 8) Patients with neurological disorders

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — their age ranged from 50-60 years
Enrollment: 40 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
. Numeric pain rating scale | up to 4 weeks
  it will measure pain intensity

SECONDARY OUTCOMES:
KOOS questionnaire | up to 4 weeks
  To measure success of range of motion
Pressure algometer | up to 4 weeks
  To measure the pain

CONTACTS AND LOCATIONS:
Locations (1):
- Kerolous Ishak Shehata Kelini, Cairo, Egypt